CLINICAL TRIAL: NCT00954863
Title: Identification and Characterization of Genotypic Resistant HIV Strains in Taiwan
Brief Title: Genotypic Resistant HIV Strains in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sui-Yuan Chang/Assistant professor, National Taiwan University
Other Study IDs: 200905045R
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-08

CONDITIONS: HIV-1; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Based on the investigators previous study, seventy-four of 786 HIV-1 isolates (9.4%), collected between 1999 to 2006, harbored one or more primary mutations associated with antiretroviral resistance to reverse-transcriptase inhibitors (RTIs) or protease inhibitors (PIs) in naïve patients. However, the drug resistance profiles for the HIV-1 integrase gene is unclear. Three objectives are proposed:

1. To investigate and compare the drug resistance profiles for the HIV-1 integrase gene between experienced and naive patients, who has not being exposed to Raltegravir.
2. To investigate and compare the drug resistance profiles for the HIV-1 integrase gene between different subtypes (subtype B, CRF01_AE and CRF07_BC).
3. To identify potential amino acid mutations in the integrase gene, which might affect the efficacy of Raltegravir.

DETAILED DESCRIPTION:
From 2008 to 2009, blood samples will be collected from consecutive HIV-1-infected patients who received HIV care at the National Taiwan University Hospital. We expect to collect 100 cases who are antiretroviral naïve and 100 cases who are treatment-experienced patients. A standardized case collection form will be used to record data of demographics and clinical characteristics and laboratory results, such as plasma HIV RNA load (PVL) and CD4 cell counts. PVL will be quantified by the Cobas Amplicor HIV-1 MonitorTM Test, version 1.5, (Roche Diagnostics Corporation, Indianapolis, USA) according to manufacturer's protocol. The CD4 cell count will be determined using FACSFlow (Becton Dickinson). This study was approved by the Institutional Review Board of the hospital.

The in-house genotypic drug resistance test will be performed to determine the drug resistance profiles for the HIV-1 pol gene, focusing on protease, reverse transcriptase, and integrase. Drug resistance mutations will be identified with the use of the HIVdb program of the Stanford University HIV Drug Resistance Database (http://hivdb.stanford.edu), in accordance with the drug-resistance mutation list of the International AIDS Society-USA Consensus Guidelines [24]. Strains with genetic mixtures of wild-type and mutant sequences at amino acid residues that code for major drug resistance will be considered to be drug resistant. Based on the interpretation given by the HIVdb program, sequences will be divided into the drug-resistant sequences, interpreted as having high, intermediate, and low levels of resistance, and the sensitive sequences, interpreted as the sensitive and potentially resistant. Multi-drug resistance (MDR) will be defined as having genotypic resistance to more than one class of antiretroviral drugs. Reference sequences of various subtypes and recombinants will be retrieved from the Los Alamos database (http://hiv-web.lanl.gov/seq-db.html). Sequences will be aligned with the Clustal W listed in the MEGA (molecular evolutionary genetics analysis) analytical package (version 3.0) [25] with minor manual adjustments. The phylogenetic trees will be constructed by the neighbor-joining method based on the Kimura 2-parameter distance matrix listed in the MEGA software. Bootstrap values greater than 750 of 1,000 replicates are considered significant.

The phenotype of those with specific or unique amino acid mutation at integrase gene will be determined using in-house phenotypic assay. Briefly, the p7 to vif fragment, about 3.6kb, will be amplified from patients' plasma viral RNA and cloned into our backbone viral clone (Figure 1). The resultant clones will be transfected into 293 cells to produce infectious viruses, whose titers will be determined by p24 assay and equal amounts of viruses will be subsequently used to infect PBMC from healthy donors. Virus titers in the supernatants from infected cells after 3, 5, and 7 days post infection in the presence or absence of tested compounds will be determined by real-time PCR or p24 assay. The minimal concentration of compounds required to reduce 50% of supernatant viral copies (EC50) will be calculated by regression analysis of the dose-response curves generated from real-time PCR or p24 assay.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals receiving clinical care at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sui-Yuan Chang, Sc. D., Principal Investigator — National Taiwan University
Locations (1):
- R424, Examination Building, National Taiwan University Hospital, Taipei, Taiwan